CLINICAL TRIAL: NCT01535768
Title: Effect of Prophylactic Aqueous Suppression on Hyperencapsulation of Ahmed Glaucoma Valves
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Credit Valley EyeCare (Industry)
Collaborators: Canadian Glaucoma Clinical Research Council (Other)
Responsible Party: Principal Investigator, Amandeep Rai, MD, Glaucoma and Advanced Anterior Segment Surgery Research Fellow, Principal Investigator, Credit Valley EyeCare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PASAGV2012
Record Dates: First submitted 2012-02-13; First posted 2012-02-20 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Timolol; dorzolamide; brinzolamide; Brimonidine Tartrate; Latanoprost; Travoprost; Bimatoprost; Acetazolamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Patients randomized to the intervention group will receive aqueous suppressant eyedrops in a stepwise fashion in order to maintain their intraocular pressure between 7-10mmHg.
  Interventions: Drug: Aqueous Suppressant Eye Drops
- Control Group (No Intervention): Patients randomized to the control group will receive standard of care treatment. They will not be aqueous suppressed within the first three postoperative months unless the bleb hyperencapsulates.
  (If they experience the hyperencapsulation phase, they will continue to receive standard of care treatment, which would then be aqueous suppressant eye drops added in a stepwise fashion)

INTERVENTIONS:
Drug: Aqueous Suppressant Eye Drops — Aqueous suppressant eye drops added stepwise to achieve IOP between 7-10mmHg. First, a beta blocker eye drop (timolol 0.25% 1 gtts in study eye BID OR timolol 0.5% 1 gtts in study eye BID).
  Next, a topical carbonic anhydrase inhibitor eye drop. (brinzolamide 1% 1 gtts in study eye TID OR dorzolamide 2% 1 gtts in study eye TID) Next, a topical alpha agonist eye drop. (brimonidine 0.1% 1 gtts in study eye TID OR brimonidine 0.15% 1 gtts in study eye TID).
  Next, a topical prostaglandin analogue eye drop. (latanoprost 0.005% 1 gtts in study eye qhs OR travoprost 0.004% 1 gtts in study eye qhs OR bimatoprost 0.01% 1 gtts in study eye qhs OR bimatoprost 0.03% 1 gtts in study eye qhs) Finally, stop the topical carbonic anhydrase inhibitor eye drop and start oral acetazolamide. (acetazolamide 250mg PO OD)
  Other Names: Timoptic; Trusopt; Azopt; Alphagan-P; Xalatan; Travatan Z; Lumigan; Diamox
  Arms: Intervention Group

SUMMARY:
After implantation of an Ahmed glaucoma valve in patients with glaucoma, hyperencapsulation phase is an unwanted postoperative phenomenon, typically occurring with the free 3 months postoperatively. When this does occur, it is treated with aqueous suppressant eye drops.

This study aims to determine if it is possible to reduce the rate of hyperencapsulation phase. Patients in the treatment group will receive aqueous suppressant eye drops before the hyperencapsulation phase starts. Treatment will be initiated once their intraocular pressure is above a pre-defined level, and will target a pre-defined range.

DETAILED DESCRIPTION:
Patients with glaucoma requiring tube shunt surgery, with or without simultaneous cataract surgery, will be enrolled in this prospective randomized controlled study at ten sites across Canada and the United States (to be determined). Patients with highly advanced glaucoma at high risk of fixation loss, neovascular glaucoma, chronic uveitis, marked corneal disease, sulfa allergy, renal disease or any contraindication to diamox use will be excluded.

Patients scheduled for Ahmed glaucoma valve surgery, with or without cataract surgery, will be randomized using a stratified central block randomization approach to the treatment group or control group. Those scheduled for combined cataract and tube shunt will be randomized separately from those receiving tube shunt alone. Surgeons will be masked to the postoperative treatment or control group at the time of surgery since randomization will occur when the patient is one-week postoperative Those in the treatment group would receive short-term prophylactic aqueous suppression for the first 3 postoperative months to maintain intraocular pressure (IOP) between 7 and 10mmHg. The control group would not receive prophylactic aqueous suppression, but would be treated using a similar protocol as the treatment group in the event that an Hyperencapsulation phase (HEP) endpoint is met.

Prophylactic aqueous suppression in the study group would only be given for the 1st 3 months postoperatively. At the 3 month visit, aqueous suppression will be stopped. The primary outcome measure is washout IOP at 4 months postoperative. Washout IOP will be checked one month after discontinuation (earlier if needed i.e., advanced glaucoma patients).

Beyond 3 months, aqueous suppressants would be used at the clinician's discretion based on IOP.

At the conclusion of the study, the 4-month postoperative washout IOP, the incidence of HEP, the 12-month IOP, the 13-month washout IOP, and medication requirement would be compared between the treatment and control arms.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of glaucoma
* scheduled for Ahmed glaucoma valve surgery, with or without simultaneous cataract surgery

Exclusion Criteria:

* neovascular glaucoma
* uveitic glaucoma
* prior tube shunt surgery
* prior cyclodestruction procedure
* abnormal cornea that would make IOP measurements unreliable
* sulfa allergy
* systemic contraindication to acetazolamide use
* inability to attend follow up visits
* intraocular pressure greater than 21 at postoperative week 1 (represents primary failure of the valve)
* anterior chamber fill within the first week postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-02; Primary Completion 2018-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 4 months postoperative
  The primary outcome measure is intraocular pressure (IOP) at 4 months postoperative. This will be a washout IOP (i.e. all glaucoma eye drops will be stopped at 3 months postoperative in all study patients)

SECONDARY OUTCOMES:
Hyperencapsulation phase (HEP) | first 3 months postoperative
  The HEP endpoint will be met within the first 3 postoperative months if all of the following are met:
  1. IOP increase by 5mmHg or greater compared to previous visit
  2. A bleb appearance in keeping with encapsulation (raised, thickened, firm, dome-shaped)
  3. no other reason for IOP increase
Qualified Ahmed Glaucoma Valve success | 12 months
  An eye will have qualified success of the Ahmed glaucoma valve if the intraocular pressure (IOP) is at or below 18mmHg at 12 months with use of medications.
Absolute Ahmed Glaucoma Valve success | 13 months
  An eye will have absolute success of the Ahmed glaucoma valve if the intraocular pressure (IOP) is at or below 18mmHg at 13 months without use of medications. Medications will be stopped at the 12 month visit, and so eyes will be washed out at 13 months.
Number of glaucoma medications | 12 months
  Will count the number of glaucoma medication classes required to achieve qualified Ahmed Glaucoma Valve success at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Devesh K Varma, MD FRCSC, Principal Investigator — University of Toronto; Ike K Ahmed, MD FRCSC, Principal Investigator — University of Toronto; Amandeep S Rai, MD, Study Director — University of Toronto
Locations (1):
- Credit Valley Eye Care, Mississauga, Ontario, Canada